CLINICAL TRIAL: NCT01440673
Title: Aprepitant for Postoperative Nausea and Vomiting in Laparoscopic Hysterectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gachon University Gil Medical Center (Other)
Collaborators: Asan Medical Center (Other); University of California, San Francisco (Other)
Responsible Party: Principal Investigator, Wol Seon Jung, Associate professor, Gachon University Gil Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: GIRBA2085
Record Dates: First submitted 2011-09-20; First posted 2011-09-26 (Estimated); Last update posted 2011-09-26 (Estimated); Status verified 2011-09

CONDITIONS: Postoperative Nausea and Vomiting
Keywords: Postoperative Nausea and Vomiting
MeSH Terms: conditions — Postoperative Nausea and Vomiting | interventions — Aprepitant

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- aprepitant 125mg (Active Comparator): NK1 receptor antagonist
  Interventions: Drug: Aprepitant
- Aprepitant 80 mg (Active Comparator)
  Interventions: Drug: Aprepitant

INTERVENTIONS:
Drug: Aprepitant — Aprepitant 80 mg, Aprepitant 125 mg

SUMMARY:
* Gynecological surgery is associated with a high incidence of postoperative nausea and vomiting.
* NK1 receptor antagonists such as aprepitant appear to be highly effective for treating acute and delayed emesis, and yet understanding of the efficacy of different doses of aprepitant is limited.
* We performed a prospective, randomized, double-blinded placebo-controlled study of 123 female adults scheduled for laparoscopic hysterectomy who received 80 mg aprepitant, 125 mg aprepitant, or a placebo.

DETAILED DESCRIPTION:
123 female patients (ages 21-60) undergoing laparoscopic hysterectomy

1. 80mg aprepitant
2. 125mg aprepitant
3. placebo

Incidences of nausea, vomiting/retching, and use of rescue antiemetics were recorded at 0, 1, 2, 24, and 48 h after surgery.

ELIGIBILITY:
Inclusion Criteria:

* female laparoscopic hysterectomy isoflurane anesthesia postoperative opioid use

Exclusion Criteria:

* liver disease neurologic disease active pulmonary disease cardiac arrhythmia allergies to any perioperative medications

Ages: 21 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 150 (Actual)
Dates: Start 2010-03; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
The numbers (and percentages) of patients who experienced complete response | 48 hours postoperatively
  * The numbers (and percentages) of patients who experienced complete response, i.e. no nausea, retching, vomiting, or need for rescue treatment
  * required rescue therapy and peak nausea scores
  * Adverse effects in the three treatment groups

CONTACTS AND LOCATIONS:
Overall Officials: WOL SEON JUNG, M.D. Ph.D., Principal Investigator — Gil Medical Center Gachon University
Locations (1):
- Gil Medical Center Gachon University, Inchon, South Korea